CLINICAL TRIAL: NCT03729479
Title: The MHERO Study (Michigan's Hypertension, Diabetes, and Obesity Education Research Online)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00146610
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Type2 Diabetes Mellitus; Hypertension; PreDiabetes; Overweight and Obesity
Keywords: dietary intervention
MeSH Terms: conditions — Hypertension; Prediabetic State; Overweight; Obesity | interventions — Dietary Approaches To Stop Hypertension; Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: 2x2 full factorial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: DASH diet (Experimental): Participants will be taught to follow a DASH diet (low-sodium and low-fat meal plan, which includes whole grains, fat-free or low-fat dairy products, vegetables, fruits, poultry, fish, and nuts, with processed, high-sodium, regular-fat, and sugar-added foods restricted).
  Interventions: Behavioral: DASH diet
- Experimental: very low carbohydrate, ketogenic diet (Experimental): Participants will be taught to follow a very low-carbohydrate, ketogenic diet (non-starchy vegetables, nuts, seeds, meat, fish, and natural fats such as avocado, olive oil, and butter, with starchy and sugary foods restricted).
  Interventions: Behavioral: Very low carbohydrate, ketogenic diet
- Experimental: DASH diet and extra support (Experimental): Participants will be taught to follow a DASH diet (low-sodium and low-fat meal plan, which includes whole grains, fat-free or low-fat dairy products, vegetables, fruits, poultry, fish, and nuts, with processed, high-sodium, regular-fat, and sugar-added foods restricted).
  They will also be given training in positive affect, mindfulness, health information seeking and sharing, and cooking practices and behavior.
  Interventions: Behavioral: DASH diet; Behavioral: Extras
- Experimental: very low carb, ketogenic diet and extra support (Experimental): Participants will be taught to follow a very low-carbohydrate, ketogenic diet (non-starchy vegetables, nuts, seeds, meat, fish, and natural fats such as avocado, olive oil, and butter, with starchy and sugary foods restricted).
  They will also be given training in positive affect, mindfulness, health information seeking and sharing, and cooking practices and behavior.
  Interventions: Behavioral: Very low carbohydrate, ketogenic diet; Behavioral: Extras

INTERVENTIONS:
Behavioral: DASH diet — Participants will be taught to follow a DASH diet (low-sodium and low-fat meal plan, which includes whole grains, fat-free or low-fat dairy products, vegetables, fruits, poultry, fish, and nuts, with processed, high-sodium, regular-fat, and sugar-added foods restricted).
  Arms: Experimental: DASH diet; Experimental: DASH diet and extra support
Behavioral: Very low carbohydrate, ketogenic diet — Participants will be taught to follow a very low-carbohydrate diet (non-starchy vegetables, nuts, seeds, meat, fish, and natural fats such as avocado, olive oil, and butter, with starchy and sugary foods restricted).
  Arms: Experimental: very low carb, ketogenic diet and extra support; Experimental: very low carbohydrate, ketogenic diet
Behavioral: Extras — Participants will be given training in positive affect, mindfulness, health information seeking and sharing, and cooking practices and behavior.
  Arms: Experimental: DASH diet and extra support; Experimental: very low carb, ketogenic diet and extra support

SUMMARY:
This study will compare the low-sodium/low-fat DASH (Dietary Approaches to Stop Hypertension) diet with a very low-carbohydrate diet, helping us to better understand how two different dietary approaches may help participants control their blood pressure, lose weight, and reduce their blood glucose.

DETAILED DESCRIPTION:
Adults with overweight or obesity, hypertension, and prediabetes or type 2 diabetes are at a high risk of adverse health outcomes including stroke, renal disease, myocardial infarction, and premature death. Evidence suggests that the first-line treatment for adults with this triple burden should be a comprehensive diet and lifestyle intervention.

However, experts disagree about which diet should be recommended. The Dietary Approaches to Stop Hypertension (DASH) diet, a lower fat diet, is the de facto diet for adults with hypertension. A very low-carbohydrate (VLC) diet, a higher fat diet, is becoming the de facto diet for weight and glycemic control. In addition, a VLC diet may reduce blood pressure through weight loss and its impact on insulin (which alters renal sodium transport and leads to diuresis). Given that these two diets, DASH and very low-carbohydrate, are extremely promising options for this population, and the fact that they have never been compared in this population or any other, this comparison is strongly warranted.

The investigators propose to use an interprofessional team (with expertise in nursing, psychology, medicine, policy, nutrition, pharmacy, and behavioral interventions) to conduct a comparative effectiveness trial of two different diets for adults with this triple burden. The HERO Study (Hypertension, Diabetes, and Obesity Education Research Online) will compare the health effects of the DASH and VLC diets.

The investigators propose one aim:

Test the feasibility, acceptability, and preliminary comparative efficacy of the interventions. The investigators will randomize 140 adults with this triple burden to the DASH or VLC versions of the 4-month intervention. Outcome measures include intervention feasibility (recruitment and retention); acceptability (satisfaction with the intervention); and preliminary comparative efficacy as determined by changes in our primary outcome (systolic blood pressure), as well as exploratory secondary outcomes (weight, glycemic control).

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 25-50
2. Diagnosis pre-hypertension or hypertension (within the past 6 months) and current resting systolic blood pressure > 130 mmHg.
3. Diagnosis of either prediabetes or type 2 diabetes, defined as:

   1. HbA1c of at least 5.7% or
   2. Two-hour glucose tolerance test >140 mg/dL
4. Aged 21-70 years old
5. Access to the internet and text messaging
6. Ability to engage in light physical activity
7. Sufficient control over their food intake to adhere to study diets
8. Willingness to regularly monitor blood pressure, glucose, dietary intake, and body weight over 4-month trial
9. Participation in the trial approved by primary care provider, along with agreement to work with the participant and our research team to manage medication changes

Exclusion Criteria:

1. Non-English speaking
2. Current use of insulin, Dilantin, lithium, and warfarin
3. Inability to complete baseline measurements
4. Severe renal or hepatic insufficiency
5. Cardiovascular dysfunction, including diagnosis of:

   1. Congestive heart failure
   2. Angina
   3. Arrhythmias
   4. Cardiomyopathy
   5. Valvular heart disease
6. Uncontrolled psychiatric disorder
7. Consumes >30 alcoholic drinks per week
8. Currently undergoing chemotherapy
9. Pregnant or planning to get pregnant in the next 12 months
10. Breastfeeding or less than 6 months' post-partum
11. Planned weight loss surgery or similar surgery performed previously
12. Vegan or vegetarian
13. Currently enrolled in a weight loss program or take weight loss supplements (that are not willing to be stopped before enrolling)
14. Expecting to move out of the area within 12 months
15. Any other medical condition that may make either diet dangerous as determined by the study medical team.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2020-08-09 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 4 months
  Measured with sphygmomanometer, assessed as change in blood pressure (systolic and diastolic blood pressure will both be measured, but systolic blood pressure is the main outcome)

SECONDARY OUTCOMES:
Glycemic control | 4 months
  Measured with HbA1c, assessed as change in HbA1c
Weight loss | 4 months
  Measured by body weight scale, assessed as change in percent body weight lost

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saslow LR, Jones LM, Sen A, Wolfson JA, Diez HL, O'Brien A, Leung CW, Bayandorian H, Daubenmier J, Missel AL, Richardson C. Comparing Very Low-Carbohydrate vs DASH Diets for Overweight or Obese Adults With Hypertension and Prediabetes or Type 2 Diabetes: A Randomized Trial. Ann Fam Med. 2023 May-Jun;21(3):256-263. doi: 10.1370/afm.2968. PMID 37217318